CLINICAL TRIAL: NCT04588467
Title: Thrombosed External Haemorrhoids During Pregnancy: Surgery Versus Conservative Treatment
Brief Title: Treatment of Thrombosed Haemorrhoids in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Russian Society of Colorectal Surgeons (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6835447
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Haemorrhoidal Crisis; Pregnancy Related
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative group (Active Comparator): Conservative treatment included dietary modification (intake of at lest 3 liters of water), stool-softeners (a 25 ml solution containing: Macrogol 3350: 13.125 g Sodium chloride: 0.3508 g Sodium hydrogen carbonate: 0.1786 g Potassium chloride: 0.0502 g) and local anesthetics application (Lidocaine 2.5%+Prilocaine 2.5%, 2g twice a day) for 10 days
  Interventions: Other: Medical treatment
- Surgical group (Experimental): Thrombectomy and local excision of external hemorrhoids were performed with the patient in the lithotomy position under local infiltrative anesthesia with UltracainDS 1:200000 1.7ml
  Interventions: Procedure: Surgical treatment

INTERVENTIONS:
Other: Medical treatment — Pregnant women complaining thrombosed haemorrhoids will receive dietary modification (intake of at lest 3 liers of water), stool-softeners (a 25 ml solution containing: Macrogol 3350: 13.125 g Sodium chloride: 0.3508 g Sodium hydrogen carbonate: 0.1786 g Potassium chloride: 0.0502 g) and local anesthetics application
  Arms: Conservative group
Procedure: Surgical treatment — Pregnant women complaining thrombosed haemorrhoids will receive local excision or thrombectomy under local anesthesia
  Arms: Surgical group

SUMMARY:
Thrombosis of the external hemorrhoids (TEH) is one of the most frequent complain during pregnancy, particularly during the third trimester.

The paucity of the medical literature on this topic has recently been underlined in the European guidelines for hemorrhoid treatment .

The aim of this prospective study is to compare the efficacy and safety of conservative versus surgical treatment of TEH in pregnant women

DETAILED DESCRIPTION:
Thrombosis of external haemorrhoids (TEH) is a quite frequent acute condition that affects women during the pregnancy arousing great concern and impacting quality of life. TEH may present as an acute hemorrhoidal crisis with severe pain and bleeding. Up to 21.8 % of pregnant females complaining of dyschezia present with a thrombosed external haemorrhoid and during last three months, 7.8 % of pregnant females experience a TEH.

Systemic changes in women body can be related to the onset of TEH and even if haemorrhoidal thrombosis does not represent a life-threatening condition during the pregnancy, on the other hand the pain can deteriorate the emotional and physical status arousing worries which affect the health system with high costs due to several accesses to the hospital.

Treatment of TEH is mainly directed to the relief of symptoms, especially pain control. Nowadays conservative and surgical management of TEH during the pregnancy have been demonstrated both effective and safe. Nevertheless, a conservative approach is more accepted as the patient's ability to tolerate the symptoms of her condition would dictate the need for surgery.

In the common practice most patients prefer to be treated conservatively experiencing resolution of their symptoms. On the other hand excision of thrombosed external haemorrhoids results in more rapid symptom resolution, lower incidence of recurrence, and longer remission intervals.

During the pregnancy the administration of conservative medications is quite limited due to the possible side effect of such drugs on the fetus.

The aim of this prospective study is to evaluate and compare the efficacy and safety of conservative and surgical treatment in patients affected by TEH during pregnancy. With regard to surgical management, thrombectomy and local excision of external haemorrhoids were compared.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* Thrombosed external haemorrhoids
* Written consent

Exclusion Criteria:

* Inflammatory bowel disease
* Cancer
* Age lower than 18 years old

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 35 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Pain evaluation: scale | 10 days
  A scale of pain will be administered to patients
Quality of Life evaluation: questionnaire | 10 days
  A questionnaire of quality of life will be administered to patients after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Inna Tulina, Prof, Study Director — Russian Society of Colorectal Surgeons
Locations (1):
- Clinic of Colorectal and Minimally invasive surgery, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Medkova Y, Tulina I, Novikov I, Nikonov A, Ischenko A, Aleksandrov L, Altomare DF, Dezi A, Picciariello A, Tsarkov P. Thrombosed external hemorrhoids during pregnancy: surgery versus conservative treatment. Updates Surg. 2024 Apr;76(2):539-545. doi: 10.1007/s13304-023-01741-y. Epub 2023 Dec 27. PMID 38151682